CLINICAL TRIAL: NCT04457921
Title: Effects of Deep Tissue Massage on Pain and Comfort After Cesarean: A Randomized Controlled Trial
Brief Title: Deep Tissue Massage on Pain and Comfort After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, ESRA GUNEY, PhD, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/57
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2020-07

CONDITIONS: Cesarean Section; Pain, Postoperative; Massage; Comfort; Midwifery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep tissue massage (Experimental): deep tissue massage applied group
  Interventions: Other: deep tissue massage
- Standard of care (No Intervention): group without deep tissue massage

INTERVENTIONS:
Other: deep tissue massage — DTM was applied to participants in the experimental group twice (at the 10th and 22nd h) after cesarean
  Arms: Deep tissue massage

SUMMARY:
The aim of this study to determine the effect of deep tissue massage applied to the back on pain and comfort after cesarean section. Personal information form was used as data collection form, Visual Analog Scala was used to assess pain, and Postpartum Comfort Questionnaire was used to assess comfort.

DETAILED DESCRIPTION:
Material and Method

This research was conducted between May 2019 and November 2019 in Inonu University Turgut Ozal Medical Center Training and Research Hospital. When power analysis was performed, the sample size was calculated to be at least 81 women for each group (81 experiments, 81 controls). Experimental group received deep tissue massage twice at 11st and 23rd hours after cesarean section. Data collection form for experimental and control groups before the first massage; Visual Analog Scala was applied four times before and after both massages. After the second massage, both groups were re-administered. Descriptive statistics and independent t-test were used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pain severity is 45 mm or more according to the Visual Analogue Scale (VAS),
* Having a single and healthy newborn,
* Does not respond negatively to any attempt to touch like massage,
* Women whose tissue integrity is complete and healthy in the area to be massaged were included in the sample.

Exclusion Criteria:

* Those with cesarean section with general anesthesia,
* Any problems diagnosed before birth and at birth (such as oligohydramnios, preeclampsia, heart disease, diabetes, placenta previa)
* Any complications related to the mother and baby in the postpartum period (bleeding, hypertension, babies taken to the neonatal intensive care unit, etc.),
* Those who received repeat doses other than routine narcotic analgesics (0.5 mg in the first 30 minutes) were not included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
pain scores | at 11st hours cesarean section
  Visual Analog Scale: Mild pain between 0-44 mm, moderate pain between 45-74 mm, and severe pain between 75-100 mm
pain scores | at 23rd hours cesarean section
  Visual Analog Scale: Mild pain between 0-44 mm, moderate pain between 45-74 mm, and severe pain between 75-100 mm

SECONDARY OUTCOMES:
comfort scores | at 23rd hours cesarean section
  Postpartum Comfort Questionnaire: The highest score from the scale is 170, the lowest score is 34. The increase in the average score obtained from the scale indicates that the comfort level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: ESRA GUNEY, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
research results will be shared.

REFERENCES:
- [Result] Simonelli MC, Doyle LT, Columbia M, Wells PD, Benson KV, Lee CS. Effects of Connective Tissue Massage on Pain in Primiparous Women After Cesarean Birth. J Obstet Gynecol Neonatal Nurs. 2018 Sep;47(5):591-601. doi: 10.1016/j.jogn.2018.07.006. Epub 2018 Aug 11. PMID 30102886
- See also: Reference link — http://pubmed.ncbi.nlm.nih.gov/30102886/
- Available data/document: Study Protocol: Mary Colleen Simonelli — http://pubmed.ncbi.nlm.nih.gov/30102886/ — web site is provided